CLINICAL TRIAL: NCT04940442
Title: Outreach and Choice in Colorectal Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Uri Ladabaum, Professor Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 61810
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-06

CONDITIONS: Colorectal Cancer Screening
MeSH Terms: interventions — Community-Institutional Relations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active choice (Experimental): FIT or colonoscopy
  Interventions: Behavioral: Outreach
- Sequential choice (Experimental): FIT offered first, then colonoscopy offered to those still unscreened
  Interventions: Behavioral: Outreach

INTERVENTIONS:
Behavioral: Outreach — Active: Outreach offering FIT or colonoscopy. Sequential: Outreach offering FIT first, and then offering colonoscopy to those still unscreened

SUMMARY:
The primary objective of this clinical trial will be to compare overall colorectal cancer (CRC) screening participation between an active choice (fecal immunochemical test [FIT] or colonoscopy) and a sequential choice (FIT offered first, then colonoscoscopy offered in those still unscreened) arm. Secondarily, we will (1) compare the proportions of FIT vs. colonoscopy per arm, (2) compare active choice vs FIT only in the initial 3 months of the study, (3) characterize changes in physician knowledge and attitudes regarding CRC screening before and after an educational seminar delivered at the launch of the initiative, (4) characterize perceptions regarding the effect of the intervention on clinical practices, and (5) compare detection rates of CRC, adenomas and SSLs per arm, and the operational results of the outreach program across arms.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 45-75 years of age not up to date with CRC screening, and without precancerous polyp history (i.e. not in post-polypectomy surveillance; ascertained based on problem list or colonoscopy results letter).
2. The assessment of screening status will happen monthly, on a rolling basis.
3. Definition of being up to date with CRC screening includes any one of the following:

   i) FIT or guaiac-FOBT within 1 year, OR

ii) Colonoscopy within 10 years, OR

iii) Sigmoidoscopy within 5 years, OR

iv) CT colonography within 5 years, OR

v) Cologuard within 3 years

Exclusion Criteria:

1. Age outside the 45-75 range.
2. History of precancerous polyps requiring colonoscopy surveillance.
3. Already being up to date with CRC screening, as defined above.
4. Evidence of total removal of the colon which would eliminate the need for screening.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with screening completion | 6 months from initial offer
  Number of patients with FIT or colonoscopy completed

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Primary Care Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No